CLINICAL TRIAL: NCT00948792
Title: The Effect of Variable Platelet Transfusion Durations on Platelet Count in Thrombocytopenic Newborns
Brief Title: Study of the Effect of Differing Platelet Transfusion Times in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Doug Dannaway / Assistant Professor of Pediatrics, University of Oklahoma Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14626
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Thrombocytopenia
Keywords: platelets; transfusion; thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long transfusion group (Active Comparator): This group of thrombocytopenic neonates who (as determined by the attending physician) are in need of a platelet transfusion will receive the transfusion over a period of two hours.
  Interventions: Procedure: Long platelet transfusion
- Short transfusion group (Experimental): This group of thrombocytopenic neonates who (as determined by the attending physician) are in need of a platelet transfusion will receive the transfusion over a period of 30 minutes.
  Interventions: Procedure: Short platelet transfusion

INTERVENTIONS:
Procedure: Short platelet transfusion — 15cc/kg of non-centrifuged, non-refrigerated, leukoreduced, AB-negative pheresis platelets administered over 30 minutes
  Arms: Short transfusion group
Procedure: Long platelet transfusion — 15cc/kg of non-centrifuged, non-refrigerated, leukoreduced, AB-negative pheresis platelets given over two hours.
  Arms: Long transfusion group

SUMMARY:
To evaluate changes in platelet counts and hemodynamics between "rapid" and "long" platelet infusion groups.

DETAILED DESCRIPTION:
1. It is our hypothesis that the change in post-transfusion platelet counts of babies who receive platelets over 30 minutes (short transfusion group) will be significantly different from the change in babies who receive platelets over two hours (long transfusion group) when platelets are checked immediately after transfusion and 6 hours after the completion of transfusion.
2. We also expect there to be significant differences in the platelet counts drawn thirty minutes after transfusion compared to the counts drawn 6 hours after the completion of the transfusion in either group.

ELIGIBILITY:
Inclusion Criteria:

* Infants with significant thrombocytopenia requiring a transfusion of platelets.

Exclusion Criteria:

* Infants requiring extracorporeal membranous oxygenation.
* Infants with congenital heart disease (other than patent foramen ovale or patent ductus arteriosus).
* Babies diagnosed with neonatal alloimmune thrombocytopenia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Dannaway, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- Children's Hospital of Oklahoma, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] British Committee for Standards in Haematology, Blood Transfusion Task Force. Guidelines for the use of platelet transfusions. Br J Haematol. 2003 Jul;122(1):10-23. doi: 10.1046/j.1365-2141.2003.04468.x. No abstract available. PMID 12823341
- [Background] Josephson CD, Su LL, Christensen RD, Hillyer CD, Castillejo MI, Emory MR, Lin Y, Hume H, Easley K, Poterjoy B, Sola-Visner M. Platelet transfusion practices among neonatologists in the United States and Canada: results of a survey. Pediatrics. 2009 Jan;123(1):278-85. doi: 10.1542/peds.2007-2850. PMID 19117893
- [Background] Murray NA, Roberts IA. Neonatal transfusion practice. Arch Dis Child Fetal Neonatal Ed. 2004 Mar;89(2):F101-7. doi: 10.1136/adc.2002.019760. PMID 14977890
- [Background] Roberts I, Murray NA. Neonatal thrombocytopenia: causes and management. Arch Dis Child Fetal Neonatal Ed. 2003 Sep;88(5):F359-64. doi: 10.1136/fn.88.5.f359. PMID 12937037
- [Background] Sola-Visner M, Saxonhouse MA, Brown RE. Neonatal thrombocytopenia: what we do and don't know. Early Hum Dev. 2008 Aug;84(8):499-506. doi: 10.1016/j.earlhumdev.2008.06.004. Epub 2008 Aug 5. PMID 18684573
- [Background] Strauss RG. How I transfuse red blood cells and platelets to infants with the anemia and thrombocytopenia of prematurity. Transfusion. 2008 Feb;48(2):209-17. doi: 10.1111/j.1537-2995.2007.01592.x. Epub 2008 Jan 7. PMID 18194380

RESULTS

PARTICIPANT FLOW:
Groups:
- Short and Long Transfusion Group: This group of thrombocytopenic neonates who (as determined by the attending physician) are in need of a platelet transfusion will receive the transfusion over a period of 30 minutes (short) or 2 hours (long).
Period: Overall Study
Arm/Group | Short and Long Transfusion Group
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Short and Long Transfusion Group: This group of thrombocytopenic neonates who (as determined by the attending physician) are in need of a platelet transfusion will receive the transfusion over a period of 30 minutes (short) or two hours (long).
Arm/Group | Short and Long Transfusion Group
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Median (Full Range); unit: Days] | 26 (.09) [1 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-transfusion Platelet Counts
Description: The difference between the baseline platelet count and the platelet count taken 30 minutes after completion of the transfusion.
Time Frame: Baseline-30 minutes after transfusion
Population: Transfusions were randomized, not babies. Therefore, each baby could provide transfusions falling into either arm of randomization. The 21 long transfusions were provided by 14 infants; the 22 short transfusions by 15. This explains the perceived discrepancy.
Measure: Median (Full Range); unit: Platelets (*10^3/mm^3)
Units Other Than Participants: transfusions
Arm/Group | Long Transfusion Group | Short Transfusion Group
Number analyzed (Participants) | 14 | 15
Number analyzed (transfusions) | 21 | 22
Platelets (*10^3/mm^3) | 99 [-19 to 442] | 97.5 [19 to 260]
Statistical Analysis 1: Comparison: Long Transfusion Group vs Short Transfusion Group; The null hypothesis is that there would be no difference in post-transfusion platelet counts (30-minutes post-transfusion) between the two groups. We opted to determine the number of transfusions that would be required to detect difference of 20,000 platelets/mm3 (with a standard deviation of 20,000). The number shown to demonstrate this was 44; Test type: Superiority or Other; p = 0.8, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Post-transfusion Platelet Counts
Description: The difference between the baseline platelet count and the platelet count taken 6 hours after completion of the transfusion.
Time Frame: Baseline - 6 hours after transfusion
Population: as for outcome 1
Measure: Median (Full Range); unit: Platelets (*10^3/mm^3)
Units Other Than Participants: Transfusions
Arm/Group | Long Transfusion Group | Short Transfusion Group
Number analyzed (Participants) | 14 | 15
Number analyzed (Transfusions) | 21 | 22
Platelets (*10^3/mm^3) | 75 [-17 to 316] | 104 [4 to 294]
Statistical Analysis 1: Comparison: Long Transfusion Group vs Short Transfusion Group; The null hypothesis is that there would be no difference in post-transfusion platelet counts (6-hour post-transfusion) between the two groups. We opted to determine the number of transfusions that would be required to detect difference of 20,000 platelets/mm3 (with a standard deviation of 20,000). The number shown to demonstrate this was 44; Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney)

3. Primary Outcome: 30 Minute-6 Hour Difference in Platelet Counts
Time Frame: 30 minutes - 6 hours after transfusion
Population: as for outcome 1
Measure: Median (Full Range); unit: Platelets (*10^3/mm^3)
Units Other Than Participants: Transfusions
Arm/Group | Long Transfusion Group | Short Transfusion Group
Number analyzed (Participants) | 14 | 15
Number analyzed (Transfusions) | 21 | 22
Platelets (*10^3/mm^3) | -17.5 [-110 to 29] | -3 [-84 to 81]
Statistical Analysis 1: Comparison: Long Transfusion Group vs Short Transfusion Group; The null hypothesis is that there would be no difference in the change in post-transfusion platelet counts (30 minutes and 6 hours post-transfusion) between the two groups. We opted to determine the number of transfusions that would be required to detect difference of 20,000 platelets/mm3 (with a standard deviation of 20,000). The number shown to demonstrate this was 44; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Transfusions were randomized, not babies. Therefore, each baby could provide transfusions falling into either arm of randomization. The 21 long transfusions were provided by 14 infants; the 22 short transfusions by 15. This explains the perceived discrepancy.
Arm/Group | Long Transfusion Group | Short Transfusion Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No